CLINICAL TRIAL: NCT04387084
Title: Short-Term Fasting Prior to Standard Checkpoint Blockade Using PD-1/PD-L1 Inhibition: A Pilot Safety and Feasibility Study
Brief Title: Short-term Fasting Prior to PD-1/PD-L1 Inhibitor Therapy for of Advanced or Metastatic Skin Malignancy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0S-20-1; NCI-2020-01590 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-20-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Advanced Malignant Skin Neoplasm; Metastatic Malignant Skin Neoplasm
MeSH Terms: conditions — Skin Neoplasms | interventions — atezolizumab; avelumab; cemiplimab; durvalumab; Immunoglobulin G; Disulfides; Nivolumab; pembrolizumab; dostarlimab; toripalimab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (STF, PD-1/PD-L1 inhibitor) (Experimental): Patients undergo STF for 47-48 hours prior to immunotherapy and for 24 hours after immunotherapy with standard of care pembrolizumab given IV over 30 minutes, nivolumab IV over 30 minutes, cemiplimab IV over 30 minutes, dostarlimab IV over 30 minutes, retifanlimab IV over 30 minutes, toripalimab IV over 60 minutes, 30 minutes for subsequent dose, tislelizumab IV over 60 minutes for 1st dose, 30 minutes for subsequent doses, avelumab IV over 60 minutes, atezolizumab IV over 60 minutes, or durvalumab IV over 60 minutes on day 3. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Avelumab; Biological: Cemiplimab; Biological: Durvalumab; Biological: Nivolumab; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Other: Short-Term Fasting; Biological: Dostarlimab; Biological: Retifanlimab; Biological: Toripalimab; Biological: Tislelizumab

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN2810
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Short-Term Fasting — Undergo STF
  Other Names: Intermittent Fasting; Short-term Intermittent Fasting
Biological: Dostarlimab — Given IV
  Other Names: Jemperli; dostarlimab-gxly
Biological: Retifanlimab — Given IV
  Other Names: Zynyz; retifanlimab-dlwr; MGA012; INCMGA-00012; INCMGA00012
Biological: Toripalimab — Given IV
  Other Names: Loqtorzi; toripalimab-tpzi; Tuoyi; ZYTORVI; JS001; TAB001; TAB-001; CHS-007; SO-001
Biological: Tislelizumab — Given IV
  Other Names: Tevimbra; tislelizumab-jsgr; BGB-A317

SUMMARY:
This trial studies the side effects of short-term fasting in patients with skin malignancy that has spread to other places in the body (advanced or metastatic) treated with a PD-L1 or PD-1 inhibitor. Immunotherapy with monoclonal antibodies, such as pembrolizumab, nivolumab, cemiplimab, avelumab, atezolizumab, or durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Undergoing short-term fasting prior to treatment with one of these PD-L1 or PD-1 inhibitors may potentially reduce the side effects of immunotherapy or even improve the effectiveness of immunotherapy in patients with skin malignancy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and feasibility of short term fasting in combination with PD-1 inhibition therapy for patients with advanced malignancy.

Ia. To estimate the percentage of patients who adhere completely to short term fasting (STF) in combination with PD-1 inhibition therapy for 3 cycles.

Ib. To estimate the percentage of patients who develop unacceptable fasting-related toxicity.

SECONDARY OBJECTIVES:

I. To measure how many patients can adhere with STF for at least 2 cycles in combination with PD-1 inhibition.

Ia. To estimate the percentage of patients who adhere to STF in combination with PD-1 inhibition therapy for at least 2 cycles, or a total of at least 6 out of 9 days.

II. To measure all grades of fasting-related toxicity. IIa. To estimate the percentage of patients who develop any grades of fasting-related toxicity, including acceptable fasting-related toxicity.

EXPLORATORY OBJECTIVES:

I. The efficacy of combining STF with PD-1/PD-L1 inhibition will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 response rate, as measured at the time of tumor assessment after 3 cycles of treatment.

II. The immune-related toxicity of combining STF with PD-1/PD-L1 inhibition will be recorded at the start of each cycle, and graded per Common Terminology Criteria for Adverse Events (CTCAE) v 4.0.

III. Quality of life during STF combined with PD-1/PD-L1 inhibition will be recorded using the Functional Assessment of Cancer Therapy - General (FACT-G) version 4, questionnaire tool.

IV. Fasting-related biomarkers to measure the impact of STF during PD-1/PD-L1 inhibition include measurement of serum insulin/IGF-1, PI3K/AKT/mTOR signaling, MAPK pathway signaling, and markers of oxidative stress.

V. Immune biomarkers will be analyzed using immunohistochemistry and ribonucleic acid (RNA) expression studies.

OUTLINE:

Patients undergo STF for 47-48 hours prior to immunotherapy and for 24 hours after immunotherapy with standard of care pembrolizumab given intravenously (IV) over 30 minutes, nivolumab IV over 30 minutes, cemiplimab IV over 30 minutes, avelumab IV over 60 minutes, atezolizumab IV over 60 minutes, or durvalumab IV over 60 minutes on day 3. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up in 3-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor malignancy for which PD-1/PDL1 inhibition based immunotherapy is recommended as standard of care therapy, as monotherapy or in combination with other checkpoint inhibitors. Acceptable PD-1/PD-L1 inhibitors include*:
* Pembrolizumab
* Nivolumab
* Cemiplimab
* Dostarlimab
* Retifanlimab
* Toripalimab
* Tislelizumab
* Atezolizumab
* Avelumab
* Durvalumab * Additional PD-1/PD-L1 inhibitors may be considered, with the approval of the principal investigator (PI), and will require a future amendment to the protocol

Other immune checkpoint inhibitors (such as those targeting CTLA-4, LAG-3, etc) that may be used in combination with PD-1/PD-L1 inhibitors as standard of care therapy include**:

* Ipilimumab
* Tremelimumab
* Relatlimab

  **Additional checkpoint inhibitors may be considered, with the approval of the PI, and will require a future amendment to the protocol.
* Advanced or metastatic cutaneous tumor with measurable disease evaluable by RECIST criteria. Patients with other solid tumors may be eligible if they have a cutaneous metastasis amenable to biopsy (with approval of PI only)
* No more than 2 lines of prior systemic therapy (not including neoadjuvant or adjuvant therapy)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count >= 1,000/mcL
* Absolute lymphocyte count >= 500/mcL
* Hemoglobin >= 8.0 g/dL
* Platelets >= 75,000/mcl
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
* Creatinine =< 1.8 mg/dl or calculated creatinine clearance > 40 ml/min
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Body mass index (BMI) >= 18.5
* Ability to understand and the willingness to sign a written informed consent and comply with short-term fasting during study and other study-related procedures

Exclusion Criteria:

* Patients with history of diabetes mellitus are not eligible for this study

  * Note: patients with pre-diabetes or a history of diabetes which subsequently resolves, who are not taking metformin or any other diabetes medications are eligible
* Patients with recent significant or unexplained weight loss that the investigator feels may pose an unacceptable risk for enrollment should be excluded. (Candidates who are overweight and have intentionally lost weight via diet or exercise should be excluded, for instance)
* Subjects on medications that may not be safely stopped during the fasting portion of the study, or which may not be safely consumed without food
* Prior history of syncope with caloric restriction in the past or other medical comorbidity which would make fasting potentially dangerous
* Prior treatment with any agent that blocks the PD-1 or PD-L1 pathway
* Prior treatment with other immune modulating agents within fewer than 4 weeks, prior to the first dose of PD-1/PD-L1 inhibition. Examples of immune modulating agents include blockers of CTLA-4, 4-1BB, OX-40, therapeutic vaccines, or cytokine therapies
* Patients must not be receiving other concomitant biologic therapy, hormonal therapy, chemotherapy, other anti-cancer therapy or any other investigational agents while on this protocol
* Radiation therapy, non-cytotoxic agents or investigational agents in the 4 weeks prior to the first dose of PD-1/PD-L1 inhibition
* Immunosuppressive systemic corticosteroids equivalent to prednisone 10 mg or greater in the 14 days prior to the first dose of PD-1/PD-L1 inhibition
* Any major surgery within 14 days prior to the first dose of PD-1/PD-L1 inhibition. Patients must have recovered from any major complications before registration
* Active autoimmune disease requiring systemic treatment in the past 2 years (i.e. use of disease modifying agents or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PD-1 or PD-L1 inhibitor
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Positive pregnancy test, active pregnancy or nursing/breast-feeding, due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants
* History of solid organ or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2027-08-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients completely adhering to 3 cycles of short term fasting (STF) (9 days of fasting) | Up to 3 cycles (each cycle is 21 days)
  Complete adherence will be defined as patients who adhere to STF (consumption of less than 200 kilocalorie [kCal] per 24 hours) in combination with PD-1/PD-L1 inhibition therapy for all 3 cycles of therapy (total of 9 days of fasting). Will be described with descriptive statistics.
Percentage of patients who develop unacceptable fasting-related toxicity | At the start of each cycle (prior to immunotherapy infusion), up to 3 cycles (each cycle is 21 days)
  Will be graded per Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The safety benchmark will be set at 0 subjects in the total cohort experiencing fasting-related toxicity, i.e., if even 1 patient experiences unacceptable fasting-related toxicity, the study will be discontinued.

SECONDARY OUTCOMES:
Percentage of patients who can partially adhere to 3 cycles of STF (9 days of fasting) | Up to 3 cycles (each cycle is 21 days)
  Partial adherence will be defined as patients who adhere to STF (consumption of less than 200 kCal per 24 hours) in combination with PD-1/PD-L1 inhibition therapy for at least 2 cycles of therapy, or at least 6 out of total 9 days of fasting. Will be described with descriptive statistics.
Incidence of acceptable fasting related toxicity | At the start of each cycle (prior to immunotherapy infusion), up to 3 cycles (each cycle is 21 days)
  Fasting-related toxicity is to be recorded at the start of each cycle (prior to immunotherapy infusion), and graded per CTCAE v 4.0. Incidence of adverse events related to fasting, including acceptable fasting-related toxicity, will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gino K In, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California